CLINICAL TRIAL: NCT02685865
Title: Randomized Trial Comparing Fully Covered, Self-Expanding Metal Stent and Plastic Stents for Endoscopic Ultrasound-guided Drainage of Walled-off Necrosis
Brief Title: Comparison of FCSEMS and Plastic Stents
Acronym: WON-MVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 837579
Record Dates: First submitted 2015-11-24; First posted 2016-02-19 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Infected Pancreatic Necrosis; Acute Pancreatic Fluid Collection; Pancreatic and Peripancreatic Necrosis; Pancreatic Collection; Symptomatic Pancreatic Necrosis
Keywords: pancreatic fluid collection; pancreatic necrosis; stent;
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCSEM Stent (Active Comparator): WON is first identified using EUS and punctured using a 19 gauge needle. 10 ml of fluid is aspirated and sent for gram stain and culture with sensitivities. Using a catheter-based stent delivery system with a 15mm AXIOS stent mounted onto it is inserted into the echoendoscope, and introduced into the WON cavity so that the stent lies within both the WON and enteric lumen. The stent is then deployed so that one flange of the stent is located within the WON cavity and the other flange is located within the enteric lumen.
  Interventions: Device: FCSEM Stent
- Plastic Stents (Active Comparator): WON is first identified using EUS, and punctured using a 19 gauge needle. 10 ml of the WON fluid is aspirated and sent for gram stain and culture with sensitivities. A 0.025 or 0.035 inch guidewire is inserted into the WON through the fine needle aspiration (FNA) needle. A transmural tract is created using an Endoscopic Retrograde Cholangiopancreatography(ERCP) catheter (with the use of a needle knife catheter ± cautery if needed), and then dilated using a 12-13.5-15mm Controlled Radial Expansion (CRE) balloon to a maximum size of 15mm if technically possible. Two or three 7 French plastic stents are inserted through the transmural tract into the WON cavity.
  Interventions: Device: Plastic Stent

INTERVENTIONS:
Device: FCSEM Stent — Hot Axios Fully covered self-expandable metal stent - Boston Scientific
  Other Names: Fully covered self-expandable metal stent
  Arms: FCSEM Stent
Device: Plastic Stent — 7 French 4 cm double pigtail plastic stent - Cook 7 French 4 cm double pigtail plastic stent - Boston Scientific
  Arms: Plastic Stents

SUMMARY:
The research design is a randomized prospective clinical trial comparing Endoscopic ultrasound (EUS) guided drainage of WON using FCSEMS and plastic stents. The trial will be conducted at the Florida Hospital Center for Interventional Endoscopy, Orlando, Florida.

DETAILED DESCRIPTION:
The research design is a randomized prospective clinical trial comparing EUS-guided drainage of WON using FCSEMS and plastic stents. The trial will be conducted at the Florida Hospital Center for Interventional Endoscopy, Orlando, Florida.The sample size estimated for this study is 60 patients. All patients will undergo EUS-guided drainage of WON and be randomized to either FCSEM or plastic stents in a 1:1 ratio using a computer-generated randomized sequence. It will not be possible to blind the endoscopist to the stent type being inserted due to the differences in stent appearance. The statistician will be blinded to the stent type utilized.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (or when applicable the subject's LAR) is capable of understanding and complying with protocol requirements.
2. The subject (or when applicable the subject's LAR) is able to understand and willing to sign an informed consent form prior to the initiation of any study procedures.
3. Males or females ≥ 18 years of age.
4. WON diagnosed on contrast-enhanced dual phase CT abdomen/pelvis (CECT) or MRI with gadolinium (seen as a fluid collection in the setting of documented pancreatic necrosis that contains necrotic material and encased within a well-defined tissue layer).
5. WON of any size with any quantity of solid/necrotic component and any no. of loculations, located within the pancreatic/peri-pancreatic space not requiring percutaneous drainage, within 2cm of the enteric wall
6. Suspected/confirmed infected WON (defined as temp ≥ 100.5°F, serum White Blood Cells ≥ 15x109/L, positive blood cultures or positive Gram stain/culture of aspirated necrotic material), and/or symptomatic WON (defined as abdominal pain, gastric/intestinal/biliary outlet obstruction resulting in nausea, vomiting, early satiety, jaundice, or persistent malaise) ≥ 4 weeks from attack of acute pancreatitis.
7. Documented history of acute or chronic pancreatitis:

   i. Acute pancreatitis is diagnosed if 2 of the following 3 criteria are met:
   1. Abdominal pain characteristic of acute pancreatitis
   2. Serum lipase/amylase ≥ x3 upper limit of normal
   3. Characteristic radiological findings of acute pancreatitis on CECT/MRI/US abdomen, such as homogeneous enhancement of pancreatic parenchyma, standing of peripancreatic fat ii. Chronic pancreatitis is diagnosed if characteristic radiological changes are seen on CT/MRI with Magnetic resonance cholangiopancreatography (MRCP) (such as pancreatic atrophy, dilated pancreatic duct, pancreatic calcification) or EUS (≥5/9 of Rosement criteria)
8. Able to undergo general anesthesia

Exclusion Criteria:

1. Females who are pregnant or lactating. Pregnancy for females of childbearing potential will be determined by routine preoperative urine or serum Human Chorionic Gonadotropin testing.
2. Irreversible coagulopathy (INR >1.5, thrombocytopenia with platelet count <50,000/mL)
3. Has surgically altered gastrointestinal anatomy such as but not limited to Billroth II, Roux-en-Y, gastric bypass
4. Age < 18 years
5. Unable to obtain consent for the procedure from either the patient or LAR
6. Use of anticoagulants that cannot be discontinued for the procedure
7. Unable to tolerate general anesthesia
8. WON that is not accessible for EUS-guided drainage
9. Percutaneous drainage of WON is required or performed prior to EUS-guided drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The number of interventions performed between metal and plastic stent groups to achieve treatment success | 6 weeks
  The primary objective of this study is to compare the number of interventions performed between metal and plastic stent groups to achieve treatment success at 6 week follow-up. Re-intervention is defined as the need for repeat EUS-guided drainage of WON using the same stent type and/or DEN and/or insertion of percutaneous catheter due to inadequate treatment response following initial WON drainage. As FCSEMS have larger diameter than plastic stents, the investigators hypothesize that the no. of re-interventions performed will be lower in the FCSEMS group compared to the plastic stent group.

SECONDARY OUTCOMES:
Technical success | at index treatment Day 0
  Successful deployment of transmural stents in to the WON cavity.
Treatment success | 6 week
  Resolution of WON on CT scan and resolution of symptoms at 6-week outpatient follow-up (from day of hospital discharge) WITHOUT the need for cross-over to minimally invasive surgical debridement
Treatment failure | 6 months
  Need for minimally-invasive surgical debridement as a consequence of inadequate endoscopic treatment response, or death as a direct consequence of WON drainage or underlying diseaseor underlying disease.
Recurrence | 6 months
  Development of WON or additional Pancreatic Fluid Collection and recurrence of symptoms following initial treatment success
Procedure duration (minutes) | at index treatment Day 0
  Time from start of the procedure (endoscope inserted into the gastrointestinal lumen to perform transmural drainage to the end of the procedure (removal of the echoendoscope/ gastroscope/ duodenoscope from the oropharynx).
Adverse events | 6 months
  Adverse event directly resulting from performing endoscopic drainage procedure. The severity will be graded according to a previously published consensus.
Duration of hospitalization | 6 months
  Day of procedure to the day of hospital discharge
Cost Analysis (Inpatient and outpatient costs) | 6 months
  Inpatient and outpatient costs of care will be calculated based on Medicare reimbursement fee structure.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — Florida Hospital Orlando
Locations (2):
- United States (2):
  - Center for Interventional Endoscopy - Florida Hospital Orlando, Orlando, Florida
  - Florida Hospital Center for Interventional Endoscopy, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] van Brunschot S, Bakker OJ, Besselink MG, Bollen TL, Fockens P, Gooszen HG, van Santvoort HC; Dutch Pancreatitis Study Group. Treatment of necrotizing pancreatitis. Clin Gastroenterol Hepatol. 2012 Nov;10(11):1190-201. doi: 10.1016/j.cgh.2012.05.005. Epub 2012 May 18. PMID 22610008
- [Background] Gardner TB, Chahal P, Papachristou GI, Vege SS, Petersen BT, Gostout CJ, Topazian MD, Takahashi N, Sarr MG, Baron TH. A comparison of direct endoscopic necrosectomy with transmural endoscopic drainage for the treatment of walled-off pancreatic necrosis. Gastrointest Endosc. 2009 May;69(6):1085-94. doi: 10.1016/j.gie.2008.06.061. Epub 2009 Feb 24. PMID 19243764
- [Background] Varadarajulu S, Bang JY, Phadnis MA, Christein JD, Wilcox CM. Endoscopic transmural drainage of peripancreatic fluid collections: outcomes and predictors of treatment success in 211 consecutive patients. J Gastrointest Surg. 2011 Nov;15(11):2080-8. doi: 10.1007/s11605-011-1621-8. Epub 2011 Jul 23. PMID 21786063
- [Background] Will U, Wanzar C, Gerlach R, Meyer F. Interventional ultrasound-guided procedures in pancreatic pseudocysts, abscesses and infected necroses - treatment algorithm in a large single-center study. Ultraschall Med. 2011 Apr;32(2):176-83. doi: 10.1055/s-0029-1245949. Epub 2011 Jan 21. PMID 21259182
- [Background] Seifert H, Biermer M, Schmitt W, Jurgensen C, Will U, Gerlach R, Kreitmair C, Meining A, Wehrmann T, Rosch T. Transluminal endoscopic necrosectomy after acute pancreatitis: a multicentre study with long-term follow-up (the GEPARD Study). Gut. 2009 Sep;58(9):1260-6. doi: 10.1136/gut.2008.163733. Epub 2009 Mar 11. PMID 19282306
- [Background] Belle S, Collet P, Post S, Kaehler G. Temporary cystogastrostomy with self-expanding metallic stents for pancreatic necrosis. Endoscopy. 2010 Jun;42(6):493-5. doi: 10.1055/s-0029-1244021. Epub 2010 Apr 29. PMID 20432209
- [Background] Berzosa M, Maheshwari S, Patel KK, Shaib YH. Single-step endoscopic ultrasonography-guided drainage of peripancreatic fluid collections with a single self-expandable metal stent and standard linear echoendoscope. Endoscopy. 2012 May;44(5):543-7. doi: 10.1055/s-0031-1291710. Epub 2012 Mar 9. PMID 22407382
- [Background] Yamamoto N, Isayama H, Kawakami H, Sasahira N, Hamada T, Ito Y, Takahara N, Uchino R, Miyabayashi K, Mizuno S, Kogure H, Sasaki T, Nakai Y, Kuwatani M, Hirano K, Tada M, Koike K. Preliminary report on a new, fully covered, metal stent designed for the treatment of pancreatic fluid collections. Gastrointest Endosc. 2013 May;77(5):809-14. doi: 10.1016/j.gie.2013.01.009. Epub 2013 Feb 26. PMID 23453183
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Forsmark CE. Management of chronic pancreatitis. Gastroenterology. 2013 Jun;144(6):1282-91.e3. doi: 10.1053/j.gastro.2013.02.008. PMID 23622138
- [Background] Stevens T. Update on the role of endoscopic ultrasound in chronic pancreatitis. Curr Gastroenterol Rep. 2011 Apr;13(2):117-22. doi: 10.1007/s11894-010-0167-3. PMID 21170612
- [Background] Bang JY, Holt BA, Hawes RH, Hasan MK, Arnoletti JP, Christein JD, Wilcox CM, Varadarajulu S. Outcomes after implementing a tailored endoscopic step-up approach to walled-off necrosis in acute pancreatitis. Br J Surg. 2014 Dec;101(13):1729-38. doi: 10.1002/bjs.9664. Epub 2014 Oct 21. PMID 25333872
- [Derived] Bang JY, Navaneethan U, Hasan MK, Sutton B, Hawes R, Varadarajulu S. Non-superiority of lumen-apposing metal stents over plastic stents for drainage of walled-off necrosis in a randomised trial. Gut. 2019 Jul;68(7):1200-1209. doi: 10.1136/gutjnl-2017-315335. Epub 2018 Jun 1. PMID 29858393